CLINICAL TRIAL: NCT06068881
Title: A Phase 2, Open-label, Single-Arm Clinical Trial to Investigate the Efficacy and Safety of Oral Tazemetostat for the Treatment of Adult Participants Age 18 and Over With Relapsed/Refractory Follicular Lymphoma Lacking the EZH2 Gain-of-Function (GOF) Mutation
Brief Title: A Study to Assess Efficacy and Safety of Oral Tazemetostat in Adult Participants With Relapsed/Refractory Follicular Lymphoma That Does Not Have an "EZH2 Gain-of-function" Genetic Mutation
Acronym: Mandolin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never started
Sponsor: Epizyme, Inc. (Industry)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-60200-452; 2023-508131-32-00 (Other: Epizyme)
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Follicular Lymphoma; Refractory Follicular Lymphoma
Keywords: EZH2 Gain-of-function; EZH2 GoF; Tazemetostat; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tazverik (Tazemetostat) (Experimental): 800mg tablet orally twice daily in continuous 28-day cycles
  Interventions: Drug: Tazverik (Tazemetostat)

INTERVENTIONS:
Drug: Tazverik (Tazemetostat) — Oral Tablet
  Other Names: IPN60200

SUMMARY:
The purpose of this research study is to learn about the effectiveness and safety of the study drug, tazemetostat, in adults with relapsed/refractory follicular lymphoma whose tumours do not have an "EZH2 gain-of-function" genetic mutation. Follicular lymphoma is a blood cancer. It affects white blood cells called lymphocytes. White blood cells normally help to fight infections, but when you have follicular lymphoma, the blood cells can form tumours in your body. 'Relapsed/refractory' follicular lymphoma means the disease has either not improved or is getting worse (progressing) during or after previous treatment.

Tazemetostat already has approval in the United States for the treatment of adult patients with relapsed/refractory follicular lymphoma with or without the "EZH2" mutation who have no satisfactory alternative treatment options.

This study is being conducted to better understand the effectiveness in patients whose tumours do not have an "EZH2 gain-of-function" genetic mutation and who previously received therapies commonly used in the U.S. in your body.

'Relapsed/refractory' follicular lymphoma means the disease has either not improved or is getting worse (progressing) during or after previous treatment.

Tazemetostat already has approval in the United States for the treatment of adult patients with relapsed/refractory follicular lymphoma with or without the "EZH2 gain-of-function" mutation who have no satisfactory alternative treatment options. This study is being conducted to better understand the effectiveness in patients whose tumours do not have an "EZH2" genetic mutation and who previously received therapies commonly used in the U.S.

In this study, all participants will receive the study drug. It will be taken by mouth (orally), as a tablet, twice daily. The sizes and number of tumours according to scan results will be collected as well as results of safety tests (such as physical examinations and laboratory tests).

The study consists of 4 periods:

* Screening period may take up to 4 weeks and require at least 1 visit.
* Treatment period will require 2 visits for each of the first 2 months, followed by 1 visit every month for the remainder of the first 12 months, followed by 1 visit every 3 months (except for women of childbearing potential [WOCBP], who will continue to have a pregnancy testing every month) until unacceptable toxicity, disease progression, or the start of new systemic anticancer therapy, whichever is first.
* Safety follow-up period will last for 1 month after the last dose of tazemetostat, and it will end with 1 visit or telephone call.
* Long-term follow-up period is only for participants who stop taking tazemetostat while their disease continues to respond; this period will last until disease progression, start of new cancer treatment, or death from any cause, whichever is first, and will require a visit every 3 months.

Tazemetostat will be provided to participants who tolerate it for as long as their disease does not progress.

Participants may be transferred to another study or program after about 2 years for continued treatment with tazemetostat or for long-term follow-up. Patients may withdraw consent to participate at any time.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, inclusive, at the time of signing the informed consent form
* Histologically confirmed follicular lymphoma (FL) grades 1, 2, or 3A
* Previously treated with ≥1 prior systemic chemotherapy, immunotherapy, or chemo-immunotherapy consistent with those used in a US population, including but not limited to bendamustine, obinutuzumab, rituximab plus lenalidomide. Patients with only 1 prior line of therapy should not be eligible for available combination or monotherapies
* Documented relapsed, refractory, or progressive disease (PD) after treatment with systemic therapy (refractory defined as less than PR or as PD <6 months after last dose)

  * Measurable disease as defined by Lugano Classification
  * Have provided sufficient tumour tissue block or unstained slides for EZH2 mutation and copy number gain (CNG) testing
* Wild-type EZH2 (ie, lacking GOF mutation). Note: If EZH2 GOF mutation status is known from site specific testing, WT patients can be enrolled with documentation of the testing, and additional archival tumour tissue or fresh lymph node biopsy taken before starting tazemetostat will be required for confirmatory testing of EZH2 GOF mutation status at study-specific laboratories. If EZH2 GOF mutation status is unknown, the results of central testing confirming wild-type (WT) EZH2 mutation status on an archival tumour sample, or a fresh lymph node biopsy is required before enrolment. (Archival tumour tissue collected within 15 months before the first dose is preferred, where feasible.)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate time between prior anticancer therapy and first dose of tazemetostat as follows:

  * Cytotoxic chemotherapy: At least 21 days.
  * Noncytotoxic chemotherapy (eg, small molecule inhibitor): At least 14 days.
  * Monoclonal and/or bispecific antibodies or chimeric antigen receptor (CAR) T: At least 28 days.
  * Radiotherapy: At least 6 weeks from prior radioisotope therapy; at least 12 weeks from 50% pelvic or total body irradiation.
* Adequate liver function, by all of the following criteria:

  * Total bilirubin ≤1.5 × the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome.
  * Alkaline phosphatase (ALP) (in the absence of bone disease), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤3 × ULN (≤5 × ULN if the patient has liver metastases).
* Adequate renal function: Calculated creatinine clearance ≥30 mL/minute per the Cockcroft and Gault formula

  * Adequate bone marrow function, by all of the following criteria:
  * Absolute neutrophil count (ANC) ≥1000/mm3 (≥1.0 × 109/L) if no lymphoma infiltration of bone marrow OR ANC ≥750/mm3 (≥0.75 × 109/L) with bone marrow infiltration: Without growth factor support (filgrastim or pegfilgrastim) for at least 14 days.
  * Platelets ≥75,000/mm3 (≥75 × 109/L), evaluated at least 7 days after last platelet transfusion.
  * Haemoglobin ≥9.0 g/dL, though may receive transfusion
* Adequate coagulation, by both of the following criteria (NOTE: In patients with thromboembolism risk, prophylactic anticoagulation, or antiplatelet therapy at investigator discretion, is recommended):
* International normalized ratio (INR) ≤1.5 × ULN
* Activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless on warfarin, then INR ≤3.0).
* Women of childbearing potential (WOCBP) must have 2 negative pregnancy tests (beta-human chorionic gonadotropin [β-hCG] on-site urine or serum tests with a minimum sensitivity of 25 mIU/mL or equivalent units of β-hCG) during screening. The second of these screening pregnancy tests

Exclusion Criteria:

* Grade 3b FL, mixed histology FL, or FL that has histologically transformed to DLBCL.
* Malignancies other than FL.
* Any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or myeloproliferative neoplasm (MPN)
* Any prior history of T-cell lymphoblastic lymphoma (LBL)/T-cell acute lymphoblastic leukaemia (ALL)
* Major surgery within 4 weeks before the first dose of study intervention.
* Significant cardiovascular impairment.
* Prolongation of corrected QT interval using Fridericia's formula (QTcF) to ≥480 msec at screening or history of long QT syndrome
* Venous thrombosis or pulmonary embolism within 3 months before starting tazemetostat. Note: Patients with deep vein thrombosis/pulmonary embolism greater than 3 months before treatment are eligible but recommended to receive prophylaxis
* Uncontrolled active infection requiring systemic therapy
* Active viral infection with human immunodeficiency virus (HIV)
* History of hepatitis B or C, unless they have adequate liver function as defined by inclusion criteria and are hepatitis B surface antigen negative with undetectable hepatitis B virus (HBV) DNA and/or have undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) if HCV antibody positive
* History of solid organ transplant
* Prior exposure to tazemetostat or other inhibitor(s) of EZH2
* Taking medications that are known strong CYP3A inhibitors and strong or moderate CYP3A inducers (including St. John's wort)
* Pregnant or lactating/breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2029-04-06 (Estimated); Study Completion 2029-04-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by an independent review committee (IRC) | From baseline to 4 months post last treatment (up to a maximum of 5 years)
  Defined as complete response + partial response [CR + PR]) in response-evaluable participants as assessed by a blinded independent review committee (BIRC).

SECONDARY OUTCOMES:
ORR assessed by the Investigator | From baseline to 4 months post last treatment (up to a maximum of 5 years)
The Best Overall Response (BOR) | From baseline to 4 months post last treatment (up to a maximum of 5 years)
  BOR as assessed by Investigator and by a BIRC.
Duration Of Response (DOR) | From baseline to 4 months post last treatment (up to a maximum of 5 years)
  DOR in participants with an objective response (CR or PR), as assessed by Investigator and by an IRC.
Progression-free survival (PFS) | From baseline to 4 months post last treatment (up to a maximum of 5 years)
  PFS from the date of the first dose of tazemetostat to the date of objective disease progression as assessed by Investigator and an IRC or to the death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | From baseline to 4 months post last treatment (up to a maximum of 5 years)
  DCR (CR + PR + Stable Disease (SD)) in response evaluable participants as assessed by Investigator and an IRC.
Percentage of participants who experience adverse events (AEs) | From baseline to 4 months post last treatment (up to a maximum of 5 years)
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The clinical significance will be graded by the investigator.
Percentage of Participants with clinically significant changes in laboratory parameters. | From baseline to 4 months post last treatment (up to a maximum of 5 years)
  Percentage of participants with clinically significant changes laboratory parameters (blood chemistry, hematology) will be reported. The clinical significance will be graded by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen